CLINICAL TRIAL: NCT00535327
Title: A Multicenter Study to Test Digital Breast Tomosynthesis (DBT) Compared to Full-Field Digital Mammography (FFDM) in Detecting Breast Cancer. Part 2. Women Undergoing Diagnostic Mammography
Brief Title: Test of Digital Breast Tomosynthesis vs. Regular Mammography in Detecting Breast Cancer in Women Undergoing Diagnostic Mammography
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: GE Healthcare - Kevin Horgan, GE Healthcare
Other Study IDs: GE 190-002
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Breast Cancer
Keywords: Mammography; mammogram; breast; Abnormal and normal breast tissue
MeSH Terms: conditions — Breast Neoplasms; Antisocial Personality Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Comparison of the ability of DBT and FFDM to detect breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years or older and has underwent screening mammography and is now referred for diagnostic mammography
* Able and willing to comply with study procedures, and have signed and dated the informed consent form
* Surgically sterile or postmenopausal

Exclusion Criteria:

* Pregnant or trying to become pregnant
* Has signs or symptoms of breast cancer
* Has been previously included in this study
* Has breast implants
* Has a history of breast cancer and is in active treatment
* Has breasts too large to be adequately positioned for the DBT examination

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women referred for diagnostic mammogram
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Longcore, Study Director — GE Healthcare